CLINICAL TRIAL: NCT03158207
Title: Safety and Efficacy of a Novel Facemask for Positive Pressure Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Tod A. Brown, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00047645
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia Induction Ventilation

STUDY DESIGN:
Intervention Model Description: The sequence of standard vs Warters mask will be determined by random number generator. Mask ventilation will be scored with both masks before and after the standard administration of paralytic medication. After grading mask ventilation the study intervention is complete and the remainder of surgical and anesthesia care will be based on the clinical needs and decisions of the care team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waters Mask (Experimental): All anesthesiologists and CRNAs will view an instructional video on the use of the Warters Mask.. Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).Mask ventilation will be scored before and after the standard administration of paralytic medication.
  Interventions: Device: Waters Mask
- Standard Mask (Active Comparator): Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).Mask ventilation will be scored before and after the standard administration of paralytic medication.
  Interventions: Other: Standard Mask

INTERVENTIONS:
Device: Waters Mask — All anesthesiologists and CRNAs will view an instructional video on the use of the Warters Mask. Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales).
  Arms: Waters Mask
Other: Standard Mask — Following induction of general anesthesia with the standard of care sequence of medications, each patient will then have mask ventilation performed and graded (Han and Warters Scales). Mask ventilation will be scored with both masks before and after the standard administration of paralytic medication.
  Arms: Standard Mask

SUMMARY:
Positive pressure ventilation can be life saving for patients who are hypoxic, hypercapneic or apneic. Manual ventilation with a facemask is a skill that is routinely required for emergency medical technicians, respiratory therapists, nurses and physicians. Although mask ventilation skills are routinely taught, even the most skilled and experienced anesthesiologists struggle to effectively mask-ventilate.

The effective use of a standard mask requires the simultaneous establishment of a seal between the mask and face and the lifting of the jaw. The preferred grip is referred to as the C&E technique. The C&E technique requires the index finger and thumb to form a "C" and push down on the mask to establish a seal between the mask and face. The lateral three fingers form the "E" and wrap under the jaw to provide lift. The grip required to establish the seal and jaw lift simultaneously is awkward and difficult to teach. The basic design of the standard facemask has not changed in approximately 100 years.

This study will evaluate a new mask design, Warters Mask, is based on a novel design that allows a far more ergonomic grip. The C&E technique is replaced by a more natural grip. With the Warters Mask, downward pressure with the palm of the hand centered on the mask provides the seal between the face and the mask. The other four fingers align under the jaw to provide lift.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Patients having elective surgery (designated by priority level of 5) requiring general endotracheal anesthesia.

Exclusion Criteria:

* Need for awake intubation based on standard preoperative evaluation by the attending anesthesiologist.
* Increased risk for aspiration of gastric contents due to full stomach, pregnancy, gastro-esophageal reflux disease, and/or hiatal hernia as identified during the pre-operative assessment.
* Previous tracheostomy procedure.
* Patient is cognitively incapable of providing their consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Warters Scale Score | one year
  The primary outcome will be the Warters Scale score for each mask, compared between patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tod Brown, MD, Principal Investigator — Assistant Professor
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided